CLINICAL TRIAL: NCT03718715
Title: The Interaction Between Metformin and Microbiota - the Reason for Gastrointestinal Side Effects?
Brief Title: The Interaction Between Metformin and Microbiota - the MEMO Study.
Acronym: MEMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Göteborg University (Other); Örebro University, Sweden (Other); Linkoeping University (Other Government); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Olov Rolandsson, Professor, Umeå University
Other Study IDs: MEMO
Record Dates: First submitted 2018-05-04; First posted 2018-10-24 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metformin; Gastrointestinal side effects; Microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples, Feces samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prospective cohort: All participants receive Metformin in accordance to the ordinary therapy practice. They will be part of one subject group/cohort. After onset of metformin treatment the subjects who develop gastrointestinal side effects will be compared with cases without gastrointestinal side effects.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Receiving Metformin is no study intervention. The investigators have no influence on the Metformin treatment. All participants receive Metformin provided by the health care system. The individual case determine dose and frequency of the treatment as part of the usual therapy guidelines.

SUMMARY:
Metformin has been used in Sweden since 1957, and it is recommended as first line therapy for type 2-diabetes (T2D) in national and international guidelines. However, adverse effects involving diarrhea, constipation, bloating, and abdominal pain are common which leads to discontinuation of medication or not being able to reach therapeutic doses. Here the investigators will perform a prospective study to investigate whether i) participants with T2D who experience adverse events following metformin treatment have an altered microbiota at baseline compared to participants without adverse events and ii) if the microbiota is altered in participants during onset of adverse events. The investigators hypothesis is that adverse effects associated with metformin are caused by an altered gut microbiota, either at base line or following metformin treatment. The study design is a nested case-cohort study. The investigators will recruit 600 patients and expect 200 individuals to have side effects and 400 without during a 24-month study period. Fecal samples will be collected at baseline, 2 months, and 4 months or when gastrointestinal symptoms occur. All fecal samples will be sequenced by 16s rRNA (ribosomal ribonucleic acid) sequencing to obtain a baseline microbiota profile; a subpopulation consisting of homogenous groups of participants will be in depth-analyzed using shotgun sequencing. If the hypothesis is confirmed this project may lead to bacterial therapies that will allow more patients tolerate metformin.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes (diagnosis set within the last 12 months)
* planned metformin treatment
* Age: 40 - 80 years
* Have provided written informed consent.

Exclusion criteria:

* already started treatment with Metformin
* intestinal disease incl. irritable bowel syndrome
* treatment with antibiotics in the last 3 months
* Inflammatory disorder t.ex. rheumatoid arthritis
* anemia, haemoglobinopathy
* alcohol or drug abuse
* cancer disease under treatment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed patients with type 2 diabetes without previous treatment with metformin.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
change from baseline in the fecal microbiota composition by detecting bacteria families with help of relative abundance (%) and diversity metrics | 4 months
  Faeces samples will be collected at baseline, after 2 months and after 4 months of Metformin treatment and analysed using 16S rRNA sequencing, whole genome shotgun sequencing and metagenomic analyses

SECONDARY OUTCOMES:
genetic correlation between Microbiota and gastrointestinal side effects | 4 months
  The microbiota genome and the relation to the appearance of gastrointestinal side effects will be analysed.
number of patients with gastrointestinal side effects | 4 months
  A questionnaire will be answered at baseline, after 2 and 4 months and refers to a period of 2 weeks before study visit. Six different side effects will be monitored: loss of appetite, nausea, vomiting, diarrhea, meteorism, stomach ache.
rate of gastrointestinal side effects | 4 months
  Changes in the rate of side effects using questionnaire at baseline, after 2 and 4 months.The answer possibilities are: never, one or a few times, daily, multiple times a day.
time to first appearance of gastrointestinal side effects | 4 months
  How many months till the onset of side effects during metformin treatment: depending on the time of assessment, 2 or 4 months
time to first appearance of side effects which requires dose changes in the Metformin treatment | 4 months
  Analysing changes in metformin treatment and relation to appearance of side effects
time to first appearance of side effects which requires termination of the Metformin treatment | 4 months
  Analysing length of metformin treatment and relation to appearance of side effects
correlation between microbiota and beneficial glucose lowering response | 4 months
  Plasma glucose will be analysed at baseline, after 2 and 4 months of Metformin treatment and correlated to the changes in the composition of microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Olov Rolandsson, Professor, Principal Investigator — Umeå University
Locations (1):
- Region Västerbotten, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No